CLINICAL TRIAL: NCT06324370
Title: Bioequivalence of Virgin Coconut Oil (VCO) Among Healthy Filipino Male Adults: An Exploratory Pharmacokinetic Study
Brief Title: Exploratory Pharmacokinetic Study of Virgin Coconut Oil (VCO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Nutrition Research Institute, Philippines (Other Government)
Collaborators: Ateneo de Manila University (Other); De La Salle Medical and Health Sciences Institute (Unknown)
Responsible Party: Principal Investigator, Carl Vincent D. Cabanilla, Senior Science Research Specialist, Food and Nutrition Research Institute, Philippines
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: FIERC-2022-023
Record Dates: First submitted 2023-12-14; First posted 2024-03-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Pharmacological Action
Keywords: Pharmacokinetic Study; Bioequivalence; Virgin Coconut Oil; Filipino; Philippines

STUDY DESIGN:
Intervention Model Description: This will be a two-sequence (single- and multiple-dose) pharmacokinetic study in healthy Filipino male human participants under fed conditions.
Masking Description: This will be an open-label pharmacokinetic study in healthy Filipino male human participants under fed conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Filipino male participants (18 to 45 yrs old) (Experimental): Healthy Filipino male participants 18 to 45 years old with optimum weight as related to height and body frame.
  1.2ml/kg/dose of virgin coconut oil (VCO) will be administered orally with 240 ml of water and standardized food for a single dose, and 0.6ml/kg/dose of virgin coconut oil (VCO) with 240 ml of water and standardized food twice a day for 7 days for multiple doses.
  Interventions: Dietary Supplement: Virgin Coconut Oil

INTERVENTIONS:
Dietary Supplement: Virgin Coconut Oil — Virgin Coconut Oil (VCO) will be administered with 240 mL water and standardized food during dosing periods.While the participant is standing up, each dose will be administered orally with at least 240 mL of water and standardized meal after an overnight fast of at least 10 hours on each occasion. The time of dosing will be recorded to the nearest minute in the case report form (CRF).
  No other liquid or solid food intake is permitted during this time. Fluid intake will be ad libitum 4 hours post-dose. There will be a washout interval of 7 days between the single- and multiple-dose studies.
  Participants will not be permitted to take any prescribed medication or over-the-counter products (including vitamins and herbal supplements) within 14 days prior to dosing or during the course of the study.
  Other Names: VCO

SUMMARY:
This is a balanced, open-label, single- and multiple-dose pharmacokinetic (PK) study of virgin coconut oil (VCO) among healthy Filipino male adults 18-45 years of age in Dasmariñas, Cavite. This study aims to determine the rate and extent of absorption of virgin coconut oil (VCO) administered in healthy male human study participants under fed conditions in single and multiple doses and to monitor the safety and tolerability of virgin coconut oil (VCO) following the standard protocol developed by the De La Salle Medical and Health Sciences Institute (DLSMHSI).

DETAILED DESCRIPTION:
Virgin coconut oil (VCO) will be administered with 240 ml water and standardized food on dosing periods, with a 5-day interval between the single-dose (0.6 ml/kg body weight) and the multiple-dose (1.2 ml/kg body weight divided into three doses daily) study periods. For the single-dose study, blood for PK analysis will be collected at pre-dose (-0.5 and 0 hours), then at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 14, and 24 hour/s post-dose. For the multiple-dose study, blood samples will be collected on the last day of dosing before the 2nd dose (at -0.5 and 0 hours), and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 14, and 24 hour/s post-dose. Sample collection will be continued after the last multiple dose at the following time points: 48, 72, 96, 120 and 144 hours. In addition, pre-dose blood samples will be collected daily from Day 8-12 to determine trough plasma concentrations and the approach to steady state. Blood samples will be sent to the Ateneo De Manila University (AdMU) for gas chromatography-mass spectrometry (GC-MS) analysis. Established primary and secondary endpoints for pharmacokinetics and safety and tolerability will be evaluated.

This study is necessary to establish human data on the pharmacokinetics of virgin coconut oil (VCO).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Filipino male
* 18-45 years of age
* signed written informed consent obtained
* body-mass index of ≥18.5 kilogram per meter-squared (kg/m2) and ≤ 24.9 kg/m2, with body weight not less than 50 kilogram(kg)

Exclusion Criteria:

* history of allergy and/or sensitivity to virgin coconut oil, any of its constituents, or related drugs
* positive Coronavirus Disease (COVID-19) Reverse Transcription-Polymerase Chain Reaction (RT-PCR) test
* history of anaphylaxis or angioedema
* systolic Blood Pressure (BP) of less than 90 mm Hg and/or diastolic BP of less than 60 mm Hg
* pulse rate of less than 50 beats/minute
* body weight +/-15% optimum weight as related to height and body frame
* history of tuberculosis or use of anti-tuberculosis drugs within 6 months prior to entry into study clinically significant gastrointestinal, cardiovascular, renal, hepatic, endocrine, metabolic, neurologic, psychiatric, hematological or other abnormalities, as judged by the Investigator
* history of QT prolongation (congenital or documented acquired QT prolongation) or ventricular cardiac arrhythmia, including torsades de pointes
* gastrointestinal disorders which may impair drug absorption, or other conditions which could modify the absorption of the study drug, as judged by the Investigator clinically significant deviation in the clinical chemistries (liver and renal function tests) and hematology at visit 1 which may impair assessment, as judged by the Investigator
* positive pre-study urine drug screen
* positive/reactive Hepatitis B and human immunodeficiency virus (HIV)
* use of any prescription drug within 30 days or any over-the-counter (OTC) drug within 14 days prior to and during the study inaccessibility of veins in left and right arm donation of blood (one unit or 350 mL) within 3 months prior to receiving the first dose of study medication
* subjects who cannot abstain from grapefruit, citrus fruits and food and/or beverages that contain caffeine or other xanthines
* an unusual diet, for whatever reason, e.g., low sodium diet, for two weeks prior to receiving any medication and throughout subject's participation in the study current smoker or smoking within two months prior to study enrollment
* consumption of alcohol for more than two years, or consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to dosing and during the study (one drink is equal to one unit of alcohol - one glass wine, half pint beer, and one measure/one ounce of spirit)
* participation in a clinical study within 3 months prior to visit 1
* significant illness during the 4 weeks preceding screening of the study
* having an occupation or requirement of driving a vehicle or operate a complex machinery before 21 days of taking the drug in both periods

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC0-t) | 25 days
  Area under the concentration-time curve from administration to the last observed concentration at time t hr
Pharmacokinetics (Cmax) | 25 days
  Maximum plasma concentration

SECONDARY OUTCOMES:
Pharmacokinetics (AUC0-inf) | 25 days
  Area under the concentration-time curve from time zero to infinity
Pharmacokinetics (tmax) | 25 days
  Time to Cmax
Pharmacokinetics (Kel) | 25 days
  Terminal elimination rate constant
Pharmacokinetics (t1/2) | 25 days
  Terminal half-life
Vital Signs (Systolic and Diastolic Blood Pressure) | 25 days
  This measures the force of blood against artery walls and can indicate cardiovascular health, risk of stroke, and other conditions like hypertension or hypotension.
Vital Signs (Pulse rate) | 25 days
  This measures the heart rate and rhythm, indicating the heart's health and overall circulatory system efficiency. An irregular or abnormal pulse can indicate cardiac issues or other systemic health problems.
Vital Signs (Body temperature) | 25 days
  Body temperature is a crucial indicator of metabolic and thermoregulatory function. Abnormal temperatures can indicate infections, inflammations, hormonal imbalances, or reactions to medication.
Vital Signs (Respiratory rate) | 25 days
  Observing the rate, depth, and pattern of breaths, respiration rate can reveal issues related to lung function and oxygenation and can even signal distress or anxiety.
Safety and Tolerability (Adverse events) | 25 days
  Adverse events
Post Study Evaluation (Fasting Blood Sugar Test) | 25 days
  Fasting Blood Sugar Test is a blood test that measures the blood sugar level in the body after at least 8 hours of fasting without food or water.
Post Study Evaluation (Blood Urea Nitrogen Test) | 25 days
  The blood urea nitrogen test also called the BUN test measures the urea nitrogen in the blood. It is recommended to diagnose kidney diseases.
Post Study Evaluation (Creatinine) | 25 days
  A Creatinine test checks the level of this chemical in either the blood or urine. Creatinine levels can provide an indicator of how well the kidneys are working.
Post Study Evaluation (Uric Acid) | 25 days
  Uric Acid test measures the levels of Uric Acid in the blood. Uric Acid is a nitrogenous compound that is formed as a by-product of metabolic activities and has been eliminated by the kidneys. This test is done to analyse gout and to measure the efficacy of medication that lowers Uric Acid.
Post Study Evaluation (Serum Glutamic Pyruvic Transaminase Test) | 25 days
  The Serum Glutamic Pyruvic Transaminase (SGPT) or Alanine Aminotransferase Test (ALT) assesses liver health, detecting liver damage, hepatitis, or monitoring conditions affecting the liver.
Post Study Evaluation (Serum Glutamic-oxaloacetic Transaminase Test) | 25 days
  A serum glutamic-oxaloacetic transaminase (SGOT) or aspartate aminotransferase (AST) test measures the levels of the enzyme AST in the blood to assess liver health. It is recommended in case of symptoms of the liver disorder, such as pain in the abdomen, nausea, vomiting, and yellow skin (jaundice).
Post Study Evaluation (Alkaline Phosphatase Test) | 25 days
  The Alkaline Phosphatase (ALP) test measures the Alkaline Phosphatase levels in the blood. Alkaline Phosphatase (ALP) is an enzyme that is found in various tissues throughout the body. The maximum concentrations of ALP are present in the cells of the bone and liver. Usually, raised levels of ALP are caused by liver disease or bone disorders.
Post Study Evaluation (TPAG- Total Protein, Albumin, Globulin Ratio Test) | 25 days
  A total protein and A/G ratio test is often included as part of a comprehensive metabolic panel, a test that measures proteins and other substances in the blood. It may also be used to help diagnose kidney disease, liver disease, or nutritional problems.
Post Study Evaluation (Indirect, Direct and Total Bilirubin) | 25 days
  Bilirubin test measures the levels of bilirubin in the blood. Higher than usual levels of bilirubin may indicate different types of liver or bile duct problems. Sometimes, higher bilirubin levels may be caused by an increased rate of destruction of red blood cells.
Post Study Evaluation (Lipid Profile - High-density lipoprotein, Low-density lipoprotein, Cholesterol and Triglycerides) | 25 days
  A complete cholesterol test - also called a lipid panel or lipid profile - is a blood test that can measure the amount of cholesterol and triglycerides in the blood. A cholesterol test can help determine the risk of the buildup of fatty deposits (plaques) in the arteries that can lead to narrowed or blocked arteries throughout the body (atherosclerosis). Results that fall outside the reference range, especially those above the upper normal level, may indicate the presence of disease or a need for further testing.
Post Study Evaluation (Lipase Test) | 25 days
  This test measures the amount of lipase in the blood. Lipase is an enzyme that is made by the pancreas. It helps the body digest fats. Higher levels of lipase may mean that one has a problem with the pancreas. Most often this means acute pancreatitis, or sudden inflammation of the pancreas.
Post Study Evaluation (Amylase Test) | 25 days
  Tests for amylase in blood or urine are mainly used to diagnose problems with the pancreas, including pancreatitis, which is an inflammation of the pancreas. It is also used to monitor chronic (long-term) pancreatitis.
Post Study Evaluation (Complete Blood Count with Platelet Count Test) | 25 days
  A complete blood count is a common blood test that is often part of a routine checkup. Complete blood counts can help detect a variety of disorders including infections, anemia, diseases of the immune system, and blood cancers.
Post Study Evaluation (Complete Urinalysis) | 25 days
  A urinalysis is a common test that can assess many different aspects of one's health with a urine sample. Healthcare providers often use urinalysis tests to screen for or monitor certain health conditions and to diagnose urinary tract infections.
Post Study Evaluation (Fecalysis) | 25 days
  A fecalysis is a series of tests done on a stool (feces) sample to help diagnose certain conditions affecting the digestive tract.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Vincent D. Cabanilla, Bachelor's, Principal Investigator — Department of Science and Technology-Food and Nutrition Research Institute (DOST-FNRI)
Locations (1):
- Department of Science and Technology-Food and Nutrition Research Institute (DOST-FNRI), City of Taguig, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No